CLINICAL TRIAL: NCT07177859
Title: A Multicenter, Randomized, Open-label, Active-controlled Phase III Clinical Trial Evaluating the Efficacy and Safety of NTQ5082 Capsules in the Treatment of Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: A Phase III Study of NTQ5082 Capsules in the Treatment of Paroxysmal Nocturnal Hemoglobinuria Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTQ5082-PNH-301
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NTQ5082 (Experimental): This group included 52 subjects, all of whom received NTQ5082 capsules 200mg qd administration
  Interventions: Drug: NTQ5082 capsules 200 mg
- Eculizumab (Active Comparator): This group included 26 subjects, all of whom received Eculizumab
  Interventions: Drug: Eculizumab Injection

INTERVENTIONS:
Drug: NTQ5082 capsules 200 mg — NTQ5082 capsules 200 mg
  Arms: NTQ5082
Drug: Eculizumab Injection — Eculizumab
  Arms: Eculizumab

SUMMARY:
NTQ5082 capsules are a small molecule CFB inhibitor. This study is a multicenter, randomized, open-label, active-controlled Phase III clinical trial designed to evaluate the efficacy and safety of NTQ5082 capsules in the treatment of patients with paroxysmal nocturnal hemoglobinuria.

ELIGIBILITY:
Inclusion Criteria:

- 1) Age ≥ 18 years, regardless of gender. 2) Subjects diagnosed with PNH according to the PNH diagnostic criteria in the Chinese "Guidelines for the Diagnosis and Treatment of Rare Diseases" (2019 edition), with PNH erythrocyte and/or granulocyte clone levels > 10% within 6 months prior to screening or during the screening period.

3) PNH patients who have not previously received complement inhibitor therapy. 4) Laboratory test (central laboratory) hemoglobin meets one of the following conditions: (1) The average hemoglobin value during screening period V1 and V2 (interval ≥ 7 days) is <100g/L; (2) If the subject receives red blood cell transfusion for PNH-related anemia during the screening period, the hemoglobin value at V1 must be <100g/L; 5) Blood lactate dehydrogenase (LDH) (central laboratory) is >1.5×upper limit of normal (ULN) during screening period V1 and V2 (interval ≥ 7 days);

Exclusion Criteria:

* 1) During the screening period, laboratory (local laboratory) results show bone marrow failure (reticulocyte count <100×109/L, or platelet count <30×109/L [must not have received platelet transfusion within 7 days prior to the laboratory test], or neutrophil count <0.5×109/L [must not have received short-acting granulocyte colony-stimulating factor within 14 days or long-acting granulocyte colony-stimulating factor within 28 days prior to the laboratory test]).

  2) During the screening period, laboratory (local laboratory) results show alanine aminotransferase (ALT), alkaline phosphatase (ALP), or gamma-glutamyltransferase (GGT) >3×ULN and the investigator determines that the patient is not suitable for study participation.

  3) Patients were receiving any of the following medications before screening, and the duration of treatment at a stable dose of the drug: (1) systemic glucocorticoids for less than 4 weeks; or prednisone or equivalent dose of glucocorticoids at a dose of >15 mg/day; (2) iron, vitamin B12, folic acid, or androgens for less than 4 weeks; (3) vitamin K antagonists (such as warfarin) with a stable international normalized ratio (INR) for less than 4 weeks; (4) low molecular weight heparin, oral anticoagulants (such as aspirin, rivaroxaban, edoxaban, apixaban) for less than 4 weeks; (5) erythropoietin (ESA), hypoxia-inducible factor prolyl hydroxylase inhibitors (HIF-PHI), or immunosuppressants (including but not limited to cyclosporine, tacrolimus, mycophenolate mofetil or mycophenolic acid, cyclophosphamide, methotrexate, etc.) for less than 8 weeks.

  4) Previous history of bone marrow/hematopoietic stem cell or solid organ transplantation (such as heart, lung, kidney, liver). 5) Patients with a history of splenectomy or planned surgery during the trial.

  6) Patients with a history of recurrent invasive infection with encapsulated bacteria (such as meningococci, Streptococcus pneumoniae, etc.), a history of systemic anti-tuberculosis treatment or current tuberculosis infection, or a history of active systemic bacterial, viral, or fungal infection within 14 days prior to the first administration of the investigational drug (defined as D1) (as determined by the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with hemoglobin (HB) levels ≥120 g/L on at least three of the four measurements between Weeks 18 and 24 in the absence of red blood cell (RBC) transfusions (defined as no RBC transfusions after Week 2 (D15) until Week 24 (D169)) | Weeks 18 to 24

SECONDARY OUTCOMES:
Proportion of subjects who had an increase in hemoglobin level ≥20 g/L from baseline on at least three of the four measurements between Weeks 18 and 24 in the absence of red blood cell transfusions (defined as no red blood cell transfusions after Week 2 | Weeks 18 to 24
Incidence and severity of adverse events | 24 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China